CLINICAL TRIAL: NCT04983511
Title: Electrical Epidural Stimulation Test for Detecting Epidural Catheter Reactivation in Obstetric Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor-Med Ctr Line, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 61999
Record Dates: First submitted 2021-07-20; First posted 2021-07-30 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Obstetric Pain; Anesthesia, Local
Keywords: Electrical Epidural Stimulation Test
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Patients with deactivated epidural/CSE catheters will be given electrical epidural stimulation test to detect its ability to be reactivated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrical Epidural Stimulation Test (EST) (Experimental): Postpartum women are given EST to predict epidural catheter reactivation for their subsequent procedures (i.e. tubal ligation).
  Interventions: Diagnostic Test: Electrical Epidural Stimulation Test (EST)

INTERVENTIONS:
Diagnostic Test: Electrical Epidural Stimulation Test (EST) — EST measures sensory/motor responses

SUMMARY:
Following labor, epidural or combined spinal-epidural (CSE) catheters are kept in place and deactivated. However, many women opt for procedures such as tubal ligation, which may require epidural anesthesia as a method of pain relief. Our study aims to confirm the ability to predict reactivation of epidural catheter in postpartum females through the electrical epidural stimulation test (EST) which was first described by the PI of this study approximately 20 years ago.

DETAILED DESCRIPTION:
In this study, investigators hope to investigate the ability of the electrical epidural stimulation test (EST) to predict reactivation of epidural catheter in postpartum females. The standard practice for confirming the reactivation of epidural or CSE catheters requires methods such as dosing the local anesthetic. With the EST test this will allow for the anesthesiologist to determine whether or not the epidural can be activated immediately.

ELIGIBILITY:
Inclusion Criteria:

* Females, 18 years and older
* American Society of Anesthesiologists physical status I or II
* Status post natural labor/birth process or C-section
* Has epidural or CSE catheter
* Upcoming procedure requiring epidural/CSE anesthesia for pain management

Exclusion Criteria:

* Contraindication to regional anesthesia
* Allergy or hypersensitivity to lidocaine, bupivacaine, or fentanyl
* Use of sedatives or opioids
* Abnormal vertebrae anatomy
* Neurological disorder with lumbar involvement
* Implanted electronic devices
* Did not receive epidural or CSE anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Electrical Epidural Stimulation Test | Duration of EST test (approximately 1-2 hours)
  Investigate the ability of the electrical epidural stimulation test (EST) to predict epidural catheter reactivation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carvalho JC, Khemka R, Loke J, Tsui BC. Low-dose intrathecal local anesthetic does not increase the threshold current for the epidural stimulation test: a prospective observational trial of neuraxial analgesia in labouring women. Can J Anaesth. 2015 Mar;62(3):265-70. doi: 10.1007/s12630-014-0291-x. Epub 2014 Dec 11. PMID 25501494
- [Result] Delgado C, Van Cleve W, Kent C, Dinges E, Bollag LA. Neuraxial anesthesia for postpartum tubal ligation at an academic medical center. F1000Res. 2018 Sep 26;7:1557. doi: 10.12688/f1000research.16025.1. eCollection 2018. PMID 30613393
- [Result] Tsui BC, Gupta S, Finucane B. Confirmation of epidural catheter placement using nerve stimulation. Can J Anaesth. 1998 Jul;45(7):640-4. doi: 10.1007/BF03012093. PMID 9717595